CLINICAL TRIAL: NCT01501656
Title: Epigenetic Testing for Breast Cancer Risk Stratification
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: STU 092011-047; BC103910 (Other Grant/Funding Number: Department of Defense Breast Cancer Research Program)
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — benign samples from unselected healthy control populations
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Promoter region hypermethylation of tumor suppressor genes is one the earliest molecular events in malignant transformation and is readily detectable in apparently normal benign breast epithelium adjacent to breast cancers. The investigators hypothesize that DNA methylation of certain genes occurs as a field change in benign breast tissue that is at high risk for malignant transformation, and as such, can be exploited for tissue-based breast cancer risk stratification. Additional work is required to identify new DNA methylation markers potentially useful for periareolar fine needle aspiration (RP-FNA)-based breast cancer risk stratification, to determine whether these markers are methylated more frequently in benign samples from women who develop breast cancer, to determine whether assessment of these markers is reproducible, to determine whether tamoxifen reduces DNA methylation, and to better understand the pattern of DNA methylation in benign samples from unselected healthy control populations. Each of these objectives contributes to advancement of a clinically useful RP-FNA-based breast cancer risk stratification test.

In addition, identification of genes that are preferentially methylated in estrogen receptor (ER) negative breast cancer will provide clues to the underlying biology responsible for this aggressive form of breast cancer. This knowledge may lead to the discovery of the causes of ER negative breast cancer, approaches for recognizing women at increased risk for this type of breast cancer, and approaches for reducing this risk.

This study seeks to identify patterns of DNA methylation in benign breast epithelial cells associated with an increased risk for breast cancer with a focus on ER negative breast cancer.

DETAILED DESCRIPTION:
Promoter region hypermethylation of tumor suppressor genes is one the earliest molecular events in malignant transformation and is readily detectable in apparently normal benign breast epithelium adjacent to breast cancers. We hypothesize that DNA methylation of certain genes occurs as a field change in benign breast tissue that is at high risk for malignant transformation, and as such, can be exploited for tissue-based breast cancer risk stratification. Additional work is required to identify new DNA methylation markers potentially useful for periareolar fine needle aspiration (RP-FNA)-based breast cancer risk stratification, to determine whether these markers are methylated more frequently in benign samples from women who develop breast cancer, to determine whether assessment of these markers is reproducible, to determine whether tamoxifen reduces DNA methylation, and to better understand the pattern of DNA methylation in benign samples from unselected healthy control populations. Each of these objectives contributes to advancement of a clinically useful RP-FNA-based breast cancer risk stratification test.

In addition, identification of genes that are preferentially methylated in estrogen receptor (ER) negative breast cancer will provide clues to the underlying biology responsible for this aggressive form of breast cancer. This knowledge may lead to the discovery of the causes of ER negative breast cancer, approaches for recognizing women at increased risk for this type of breast cancer, and approaches for reducing this risk.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 30 and 79.
* Untreated stage 1 - 3 invasive breast cancer or a woman never diagnosed with breast cancer.
* BI-RADS 1, 2, or 3 breast imaging within 12 months for women >40 years of age recruited into the control group.

Exclusion Criteria:

* <30 or >80 years of age
* Unable to provide informed consent
* Presence of an undefined palpable or mammographic breast lesion suspicious for malignancy (BIRADS 4 or 5)
* Breast implants
* Bilateral prophylactic mastectomy
* Any prior breasts irradiation
* Any systemic chemotherapy in the past
* Performance status that restricted normal activity for a significant portion of the day
* Use of luteinizing-hormone-releasing-hormone (LHRH) analogs, prolactin inhibitors, antiandrogens, or systemic glucocorticoids within three months
* Ever use of tamoxifen, raloxifene, or other SERMs
* Ever use of aromatase inhibitors
* Pregnancy or lactation within six months
* Bleeding diathesis of any kind

  1. Inherited coagulation disorder
  2. Current coumadin use
  3. Use of drugs that inhibit platelet aggregation within 10 days

Ages: 30 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Archived tumor tissue, Newly diagnosed primary breast cancer patients and healthy women who have never been diagnosed with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
DNA methylation | 2 years
  This objective assesses methylation of seven genes in 97 archival breast cancer samples.

SECONDARY OUTCOMES:
Frequency of methylation | 2 years
  Measure the frequency of methylation of ER positive and ER negative breast cancer-associated genes in benign breast epithelial cells obtained by RP-FNA.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Brekken, MD, Principal Investigator — UT Southwetstern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No